CLINICAL TRIAL: NCT00218374
Title: Hyperalgesia in Methadone Patients: Can it be Treated?
Brief Title: Dextromethorphan, Gabapentin, and Oxycodone to Treat Opioid-Induced Hyperalgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Margaret (Peggy) Compton, UCLA School of Nursing
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA-15463-1; R01-15463-1; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-08

CONDITIONS: Hyperalgesia; Opioid-Related Disorders
Keywords: Opiate Addiction; Opiate Dependence
MeSH Terms: conditions — Hyperalgesia; Opioid-Related Disorders | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Drug: Gabapentin — Gabapentin initiated up to a daily dose of 2400mg PO x 5 weeks

SUMMARY:
Individuals who reduce or stop use of opioid medications are at risk for developing hyperalgesia, which is an increased sensitivity to pain. This study will compare the effectiveness of dextromethorphan, gabapentin, and oxycodone at reducing hyperalgesia in individuals addicted to opioids who are concurrently receiving methadone treatment.

DETAILED DESCRIPTION:
Opioid medications are frequently used for the treatment of moderate to severe pain; however, individuals who use opioids have a high risk of becoming addicted. Opioid users who abruptly stop using opioid drugs may experience withdrawal symptoms, including drug craving, sweating, sleep disruption, nausea, irritability, and pain. Hyperalgesia, a severe and excessive sensitivity to pain, is a serious condition that may also occur when opioid use is reduced or discontinued. Opioid medications affect both the pain inhibitory and facilitatory systems, meaning that while they are effective at treating pain in many individuals, they also have the ability to intensify pain and cause hyperalgesia in some opioid users. Three medications, dextromethorphan, gabapentin, and oxycodone, may alleviate the symptoms of hyperalgesia and lessen an individual's sensitivity to pain. Further research is needed to confirm the benefits of these medications for opioid addicts. The purpose of this study is to compare the effectiveness of dextromethorphan, gabapentin, and oxycodone at reducing opioid-induced hyperalgesia in methadone-maintained opioid addicts.

This study will involve three separate experiments. Participants in Experiment 1 will be randomly assigned to receive either dextromethorphan or placebo; in Experiment 2, participants will be randomly assigned to receive either gabapentin or placebo; and in Experiment 3, participants will be randomly assigned to receive either oxycodone or placebo. Each experiment will last 5 weeks. All 3 experiments will begin with a screening session. Potential participants will undergo a physical exam and an electrocardiogram. Blood and urine will be collected for laboratory tests and drug screening. Each individual's medical and drug history will be reviewed and psychological and opiate withdrawal symptoms will be assessed. Individuals who complete the screening and meet all study requirements will be permitted to continue in the study.

All participants will be maintained on methadone throughout the study. Participants will also receive either the study medication (dextromethorphan, gabapentin, or oxycodone) or placebo four times per day beginning on Day 5. Study visits will take place once a week. At each visit, medications for the previous week will be accounted for and medications for the following week will be dispensed. Questionnaires and self-reports will be completed to assess depression levels and drug use. Urine tests will be used to screen for the presence of drugs and alcohol. During the study, participants will take part in four pain testing sessions to measure pain threshold and tolerance; two sessions will take place during Week 1 and another two sessions will occur during Week 5. The pain testing sessions will include a cold pressor (CP) test and an electrical stimulation (ES) procedure. The CP test will involve placing an arm in ice water for a short period of time; the ES procedure will involve stimulating muscle nerve endings via electrodes placed on the skin. Immediately after the CP and ES sessions, blood will be drawn for laboratory testing. Participants will again complete questionnaires and self-reports, and urine samples will be collected. Gift cards will be offered as an incentive for attending study visits and having negative drug tests.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 55 years of age.
* Meets DSM-IV diagnostic criteria for opioid dependence
* Taking a stable dose of methadone for 6 weeks prior to study entry and is compliant in methadone maintenance treatment
* Is in good physical health or under a physician's care if a medical condition requires ongoing treatment

Exclusion Criteria:

* Known sensitivity to dextromethorphan, gabapentin, or oxycodone
* Currently dependent on alcohol, benzodiazepine, or any drug (other than nicotine)
* Currently in an acutely psychotic, severely depressed state and in need of inpatient treatment
* Immediate suicide risk
* Neurological or psychiatric illness (e.g., peripheral neuropathy, schizophrenia, neuropathic pain, Raynaud's disease, or urticaria)
* Acute medical condition that would make study participation medically dangerous (e.g., acute hepatitis, unstable cardiovascular disease, liver disease, or kidney disease)
* Liver enzyme values five times greater than normal
* Currently taking analgesic medication for a painful condition on a regular basis
* Current or past history of high blood pressure, heart disease, or stroke
* Currently using a pacemaker
* Pregnant or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2006-10; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Pain response (measured after each pain testing session on Days 1, 4, 36, and 39) | 6 week

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Compton, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States